CLINICAL TRIAL: NCT03868059
Title: Ambulatory Blood Pressure Monitoring in Oral Testosterone Undecanoate (TU, LPCN 1021) Treated Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPCN 1021-18-001
Record Dates: First submitted 2019-02-21; First posted 2019-03-08 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Hypogonadism, Male
MeSH Terms: conditions — Eunuchism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LPCN 1021 (Experimental): LPCN 1021 at a 225 mg dose taken twice daily (total daily dose of 450 mg taken as 225 mg in the morning and 225 mg in the evening),
  Interventions: Drug: LPCN 1021

INTERVENTIONS:
Drug: LPCN 1021 — LPCN 1021 is gelatin capsule product provided as 112.5 mg testosterone undecanoate per capsule.
  Other Names: TLANDO

SUMMARY:
This is an open-label, multi-center, single arm study evaluating the blood pressure (BP) changes from baseline (Visit 3) to post-treatment (Visit 5) assessed by ambulatory blood pressure monitoring (ABPM) in LPCN 1021 treated adult hypogonadal male subjects.

DETAILED DESCRIPTION:
This is an open-label, multi-center, single arm study evaluating the blood pressure (BP) changes from baseline (Visit 3) to post-treatment (Visit 5) assessed by ambulatory blood pressure monitoring (ABPM) in LPCN 1021 treated adult hypogonadal male subjects.

The study is comprised of six scheduled visits: Visit 1 and 2 are for screening, Visit 3 is to assess subject's baseline BP and pulse rate (PR) via ABPM. Visit 4 is to enroll subjects, and to provide subjects with study medication for the start of dosing. Visit 5 is to assess subject's post-treatment BP and PR via ABPM. Visit 6 is to perform exit visit procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date the study consent form(s) which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
2. Male between 18 and 80 years of age, inclusive, with documented onset of hypogonadism prior to age 65.
3. Subjects should be diagnosed to be primary (congenital or acquired) or secondary hypogonadal (congenital or acquired).
4. Serum total T below lab normal range (300 ng/dL) based on two consecutive blood samples obtained between 6 and 10 AM, on two separate days at approximately the same time of day, following an appropriate washout of current androgen replacement therapy, if required.
5. Naïve to androgen replacement or has discontinued current treatment and completed adequate washout of prior androgen therapy. Washout must be completed prior to collection of baseline serum T samples to determine study eligibility.
6. Judged to be in good general health as determined by the investigator at screening.

Exclusion Criteria:

1. History of significant sensitivity or allergy to androgens, or product excipients.
2. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

   1. Hemoglobin < 11.5 g/dL or > 16.5 g/dL
   2. Hematocrit < 35% or > 54%
   3. Serum transaminases > 2.5 times upper limit of normal
   4. Serum bilirubin > 2.0 mg/dL
   5. Creatinine > 2.0 mg/dL
   6. PSA > 4 ng/mL
   7. Prolactin > 17.7 ng/mL.
3. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up.
4. Subjects with screening systolic BP or diastolic BP above 160 mmHg or 100 mmHg, respectively.
5. Subjects with symptoms of moderate to severe benign prostatic hyperplasia.
6. History of seizures or convulsions occurring after age 5, including alcohol or drug withdrawal seizures.
7. History of gastric surgery, cholecystectomy, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
8. History of any clinically significant illness, infection, or surgical procedure within 1 month prior to study drug administration.
9. Known tolerability issues with ABPM devices.
10. History of stroke, myocardial infarction, transient ischemic attack, or acute coronary syndrome within the past 5 years.
11. History of long QT syndrome (or QTcB > 450) or unexplained sudden death (including cardiac death) or history of long QT syndrome in a first degree relative (parent, sibling, or child).
12. Subjects who are not on stable dose of current medication (no changes in medication in the last 3 months).
13. History of current or suspected prostate or breast cancer.
14. History of untreated obstructive sleep apnea or not compliant with sleep apnea treatment.
15. Active alcohol or any drug substance abuse, or history of abuse that will interfere with the subject's ability to participate in the study in the judgement of the investigator.
16. Use of known inhibitors (e.g., ketoconazole) or inducers (e.g., dexamethasone, phenytoin, rifampin, carbamazepine) of cytochrome P450 3A (CYP3A) within 30 days prior to study drug administration and through the end of the study. A list of prohibited medications is provided in Appendix C.
17. Use of any investigational drug within 5 half-lives of the last dose in the past 6 months prior to Study Day -2 without principal investigator and/or sponsor approval.
18. Receipt of any investigational drug by injection within 30 days or 10 half-lives (whichever is longer) prior to study drug administration without principal investigator and/or sponsor approval.
19. Subject who is not willing to use adequate contraception for the duration of the study.
20. Any contraindications to a MRI scan (i.e. subjects with non-removable ferromagnetic implants, pacemakers, aneurysm clips or other foreign bodies), and/or subjects with claustrophobic symptoms and/or inability to fit into an MRI scanner.
21. Inability to understand and provide written informed consent for the study.
22. Considered by the investigator or the sponsor-designated physician, for any reason, that the subject is an unsuitable candidate to receive LPCN 1021 (exact reason should be specified by the investigator).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Delconte, MD, Study Director — Lipocine Inc.
Locations (16):
- United States (16):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - South Florida Medical Research, Aventura, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Neostart Corporation dba AGA Clinical Trials, Hialeah, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Regional Urology, Shreveport, Louisiana
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Aventiv Research, Inc., Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Granger Medical Clinic, West Valley City, Utah
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] White WB, Dobs A, Carson C, DelConte A, Khera M, Miner M, Shahid M, Kim K, Chidambaram N. Effects of a Novel Oral Testosterone Undecanoate on Ambulatory Blood Pressure in Hypogonadal Men. J Cardiovasc Pharmacol Ther. 2021 Nov;26(6):630-637. doi: 10.1177/10742484211027394. Epub 2021 Jun 30. PMID 34191621

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LPCN 1021
Started | 138
Completed | 126
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Safety Set - Subjects who have received at least 1 dose of study drug
Arm/Group | LPCN 1021
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 109
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 138
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.12 (5.75)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ambulatory Blood Pressure Monitoring (ABPM)-Measured Average 24-hour Systolic Blood Pressure (SBP)
Description: Change in average systolic blood pressure as measured by ambulatory blood pressure monitoring (ABPM) from Visit 3 (Baseline) to Visit 5 (End of Study)
Time Frame: Baseline to end of study (approximately 4 months).
Population: Subjects who had evaluable average 24-hour SBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 118
mmHg | 3.8 (11.8)

2. Secondary Outcome: Change in ABPM-measured Average Daytime SBP
Description: Change in average daytime SBP as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average daytime SBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
mmHg | 5.2 (14.9)

3. Secondary Outcome: Change in ABPM-measured Average Nighttime SBP
Description: Change in average nighttime SBP as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with evaluable average nighttime SBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
mmHg | 4.3 (16.7)

4. Secondary Outcome: Change in ABPM-measured Average 24-hour Diastolic Blood Pressure (DBP)
Description: Change in average 24-hour DBP as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with evaluable average 24-hour DBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 118
mmHg | 1.2 (4.9)

5. Secondary Outcome: Change in ABPM-measured Average Daytime DBP
Description: Change in average daytime DBP as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average daytime DBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
mmHg | 1.7 (6.5)

6. Secondary Outcome: Change in ABPM-measured Average Nighttime DBP
Description: Change in average nighttime DBP as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average nighttime DBP measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
mmHg | 1.7 (7.2)

7. Secondary Outcome: Change in ABPM-measured Average 24-hour Pulse Rate (PR)
Description: Change in average 24-hour pulse rate as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average 24-hour PR measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LPCN 1021
Number analyzed (Participants) | 118
bpm | 2.0 (5.9)

8. Secondary Outcome: Change in ABPM-measured Average Daytime PR
Description: Change in average daytime pulse rate as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average daytime PR measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
bpm | 2.6 (6.9)

9. Secondary Outcome: Change in ABPM-measured Average Nighttime PR
Description: Change in average nighttime pulse rate as measured by ABPM from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable average nighttime PR measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
bpm | 0.44 (7.2)

10. Secondary Outcome: Change in Morning SBP Measured in Triplicate at the Clinic
Description: Change in morning systolic blood pressure measured in triplicate at the clinic from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable morning SBP measurements in triplicate at the clinic at Baseline and end of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 127
mmHg | 4.8 (12.4)

11. Secondary Outcome: Change in Morning DBP Measured in Triplicate at the Clinic
Description: Change in morning diastolic blood pressure measured in triplicate at the clinic from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable morning DBP measurements in triplicate at the clinic at Baseline and end of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 127
mmHg | 1.6 (7.9)

12. Secondary Outcome: Change in Morning PR Measured in Triplicate at the Clinic
Description: Change in morning pulse rate measured in triplicate at the clinic from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable morning PR measurements in triplicate at the clinic at Baseline and End of Study
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LPCN 1021
Number analyzed (Participants) | 127
bpm | 2.0 (9.8)

13. Secondary Outcome: Change in Patient Reported Sexual Distress
Description: Change in patient reported sexual distress from visit 3 to Visit 5 Female Sexual Distress Scale - Revised, Item 13 Possible scores range from 0 (better) to 4 (worse)
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with evaluable patient reported sexual distress questionnaire responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LPCN 1021
Number analyzed (Participants) | 125
units on a scale | -0.3 (1.32)

14. Secondary Outcome: Change in Patient Reported Sexual Desire
Description: Change in patient reported sexual desire from visit 3 to Visit 5 Psychosexual Daily Questionnaire Possible scores range from 0 (worse) to 5 (better)
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with evaluable patient reported sexual desire questionnaire responses
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LPCN 1021
Number analyzed (Participants) | 125
units on a scale | 1.2 (1.1)

15. Secondary Outcome: Percent Relative Change in MRI-PDFF From Baseline (MRI-1) to Interim Analysis (MRI-2)- Subgroup: MRI-PDFF of ≥5%
Description: Percent Relative Change in Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) from Baseline (MRI-1) to Interim Analysis (MRI-2) in subjects with a baseline MRI-PDFF of ≥5%
Time Frame: Baseline (MRI-1) to Interim Analysis (MRI-2) (Approximately 8 Weeks)
Population: Subjects with evaluable baseline and interim MRI-PDFF data, with MRI-PDFF measurement of ≥5% at baseline
Measure: Mean (Standard Deviation); unit: % Relative Change
Arm/Group | LPCN 1021
Number analyzed (Participants) | 20
% Relative Change | -13.5 (49.0)

16. Secondary Outcome: Percent Relative Change in MRI-PDFF From Baseline (MRI-1) to Post-Treatment Analysis (MRI-3)- Subgroup: MRI-PDFF of ≥5%
Description: Percent Relative Change in Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) from Baseline (MRI-1) to Post-Treatment Analysis (MRI-3) in subjects with a baseline MRI-PDFF of ≥5%
Time Frame: Baseline (MRI-1) to Post-Treatment Analysis (MRI-3) (Approximately 16 Weeks)
Population: Subjects with evaluable baseline and post-treatment MRI-PDFF data, with MRI-PDFF measurement of ≥5% at baseline
Measure: Mean (Standard Deviation); unit: % Relative Change
Arm/Group | LPCN 1021
Number analyzed (Participants) | 21
% Relative Change | -33.4 (31.5)

17. Secondary Outcome: Percent Relative Change in MRI-PDFF From Baseline (MRI-1) to Interim Analysis (MRI-2)- Subgroup: MRI-PDFF of ≥10%
Description: Percent Relative Change in Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) from Baseline (MRI-1) to Interim Analysis (MRI-2) in subjects with a baseline MRI-PDFF of ≥10%
Time Frame: Baseline (MRI-1) to Interim Analysis (MRI-2) (Approximately 8 Weeks)
Population: Subjects with evaluable baseline and interim MRI-PDFF data, with MRI-PDFF measurement of ≥10% at baseline
Measure: Mean (Standard Deviation); unit: % Relative Change
Arm/Group | LPCN 1021
Number analyzed (Participants) | 7
% Relative Change | -38.5 (27.5)

18. Secondary Outcome: Percent Relative Change in MRI-PDFF From Baseline (MRI-1) to Post-Treatment Analysis (MRI-3)- Subgroup: MRI-PDFF of ≥10%
Description: Percent Relative Change in Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF) from Baseline (MRI-1) to Post-Treatment Analysis (MRI-3) in subjects with a baseline MRI-PDFF of ≥10%
Time Frame: Baseline (MRI-1) to Post-Treatment Analysis (MRI-3) (Approximately 16 Weeks)
Population: Subjects with evaluable baseline and post-treatment MRI-PDFF data, with MRI-PDFF measurement of ≥10% at baseline
Measure: Mean (Standard Deviation); unit: % Relative Change
Arm/Group | LPCN 1021
Number analyzed (Participants) | 8
% Relative Change | -39.7 (32.6)

19. Other Pre Specified Outcome: Change is SBP Dip
Description: Change in systolic blood pressure dip, as defined as the difference between daytime mean systolic blood pressure and nighttime mean systolic blood pressure, from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects who had evaluable SBP dip measurements from Baseline to End of Study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 126
mmHg | 0.5 (9.4)

20. Other Pre Specified Outcome: Change in ABPM-measured Average 24-hour SBP in Subjects With a Low Framingham Risk Score (FRS)
Description: Change in average 24-hour SBP in subjects with a low cardiovascular risk based on their Framingham Risk Score (0<FRS<11) from Visit 3 (Baseline) to Visit 5 (End of Study); Risk Level: Low: 0<FRS<11; Moderate: 11≤FRS<24; High: FRS≥24.
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with a low FRS (0<FRS<11) who had evaluable 24-hour SBP measurements from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 40
mmHg | 2.6 (2.7)

21. Other Pre Specified Outcome: Change in ABPM-measured Average 24-hour SBP in Subjects With a Moderate Framingham Risk Score (FRS)
Description: Change in average 24-hour SBP in subjects with a moderate cardiovascular risk based on their Framingham Risk Score (11≤FRS<24) from Visit 3 (Baseline) to Visit 5 (End of Study); Risk Level: Low: 0<FRS<11; Moderate: 11≤FRS<24; High: FRS≥24.
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with a medium FRS (11≤FRS<24) who had evaluable 24-hour SBP measurements from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 74
mmHg | 4.8 (13.1)

22. Other Pre Specified Outcome: Change in ABPM-measured Average 24-hour SBP in Subjects With a High Framingham Risk Score (FRS)
Description: Change in average 24-hour SBP in subjects with a high cardiovascular risk based on their Framingham Risk Score (FRS≥24) from Visit 3 (Baseline) to Visit 5 (End of Study); Risk Level: Low: 0<FRS<11; Moderate: 11≤FRS<24; High: FRS≥24.
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with a high FRS (FRS≥24) who had evaluable 24-hour SBP measurements from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 4
mmHg | -1.8 (14.9)

23. Other Pre Specified Outcome: Change in ABPM-measured Average 24-hour SBP in Subjects With a Baseline SBP >140mmHg
Description: Change in average 24-hour SBP as measured by ABPM in subjects with a baseline SBP >140mmHg from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with a baseline SBP >140mmHg who had evaluable average 24-hour SBP measurements from baseline to end of study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LPCN 1021
Number analyzed (Participants) | 25
mmHg | -3.0 (13.7)

24. Other Pre Specified Outcome: Change in Hematocrit From Baseline
Description: Change in Hematocrit (%) from Visit 3 to Visit 5
Time Frame: Baseline to end of Study (approximately 4 months)
Population: Subjects with evaluable Hematocrit values from baseline and end of study
Measure: Mean (Standard Deviation); unit: percentage of hematocrit
Arm/Group | LPCN 1021
Number analyzed (Participants) | 129
percentage of hematocrit | 3.2 (3.6)

25. Other Pre Specified Outcome: Number of Participants Who Started a New Hypertensive Medication or Increased Their Hypertensive Medication Dose
Description: Number of participants who had to start a new hypertensive medication or increase their hypertensive medication dose from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | LPCN 1021
Number analyzed (Participants) | 138
Participants | 2

26. Other Pre Specified Outcome: Change in Hemoglobin From Baseline
Description: Change in Hemoglobin from Visit 3 to Visit 5
Time Frame: Baseline to End of Study (approximately 4 months)
Population: Subjects with evaluable Hemoglobin values from baseline and end of study
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LPCN 1021
Number analyzed (Participants) | 129
g/dL | 0.87 (1.05)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | LPCN 1021
All-Cause Mortality (participants affected / at risk) | 0/138
Serious Adverse Events (participants affected / at risk) | 2/138
Other Adverse Events (participants affected / at risk) | 22/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPCN 1021 (N=138)
Psychiatric Disorders (Psychiatric disorders) | 1 — Schizoaffective Disorder Bipolar Type
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 1 — Arthritis
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LPCN 1021 (N=138)
Polycythemia (Blood and lymphatic system disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (7)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2)
Haematocrit increased (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT03868059/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT03868059/SAP_001.pdf